CLINICAL TRIAL: NCT03329846
Title: A Phase 3, Randomized, Double-blind Study of BMS-986205 Combined With Nivolumab Versus Nivolumab in Participants With Metastatic or Unresectable Melanoma That is Previously Untreated
Brief Title: An Investigational Immuno-therapy Study of BMS-986205 Combined With Nivolumab, Compared to Nivolumab by Itself, in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA017-055; 2017-002499-14 (EudraCT Number)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — linrodostat; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Placebo (Active Comparator): Specified dose on specified day
  Participants will no longer receive BMS-986205 Placebo
  Interventions: Biological: Nivolumab; Drug: Placebo
- Nivolumab + BMS-986205 (Experimental): Specified dose on specified day.
  Participants have the option to discontinue BMS-986205, and continue nivolumab monotherapy, at investigator discretion
  Interventions: Drug: BMS-986205; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986205 — specified dose on specified day
  Arms: Nivolumab + BMS-986205
Biological: Nivolumab — Specified dose on specified day
  Other Names: BMS-936558
Drug: Placebo — Specified dose on specified day
  Other Names: BMS-986205 matching placebo
  Arms: Nivolumab + Placebo

SUMMARY:
The purpose of this study is to see if BMS-986205 combined with nivolumab, compared to nivolumab by itself, is more effective in treating Melanoma that has spread or is unable to be removed by surgery, and has not previously been treated

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* 12 years and older unless not permitted by local regulations; in that case 18 years old and older
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1
* Histologically confirmed Stage III (unresectable) or Stage IV melanoma, per the American Joint Committee on Cancer (AJCC) Staging Manual (8th edition)
* Treatment-naïve participants (no prior systemic anticancer therapy for unresectable or metastatic melanoma)
* Measurable disease per RECIST v1.1

Exclusion Criteria:

* Active brain metastases or leptomeningeal metastases
* Uveal or ocular melanoma
* Participants with active, known, or suspected autoimmune disease
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (60):
- United States (6):
  - Angeles Clinic and Research Institute, Los Angeles, California
  - University Of Colorado, Aurora, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University Of Chicago, Chicago, Illinois
  - Oregon Health & Science University, Portland, Oregon
  - Local Institution, Seattle, Washington
- Australia (6):
  - Local Institution, Blacktown, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Box Hill, Victoria
  - Local Institution, Melbourne, Victoria
- Canada (2):
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Czechia (3):
  - Klinika onkologie a radioterapie, Hradec Králové
  - Dermatovenerologicka klinika 3. LF UK a FNKV, Prague
  - Dermatovenerologicka klinika VFN a 1. LF UK, Prague
- France (3):
  - Local Institution, Boulogne-Billancourt
  - Local Institution, Saint-Etienne
  - Local Institution, Villejuif
- Germany (9):
  - Elbe Klinikum Buxtehude, Buxtehude
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Local Institution, Essen
  - SRH Wald-Kliniken Gera GmbH, Gera
  - Georg August Universitaet Goettingen, Göttingen
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, München
  - Local Institution, Tübingen
- Interbalkan European Medical Center, Thessaloniki, Greece
- Ireland (2):
  - Local Institution, Dooradoyle, Limerick
  - Local Institution, Dublin
- Italy (3):
  - Local Institution, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Azienda Ospedaliera Universitaria Senese, Siena
- Japan (5):
  - Local Institution, Sendai, Miyagi
  - Local Institution, Niigata, Niigata
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Chuo-ku, Tokyo
- Netherlands (4):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
- New Zealand (2):
  - Local Institution, Christchurch
  - Local Institution, Wellington
- Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw, Poland
- Spain (6):
  - Local Institution, Barcelona
  - Local Institution, Jaén
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Santiago Compostela
  - Local Institution, Valencia
- Universitaetsspital Zuerich, Zurich, Switzerland
- United Kingdom (6):
  - Local Institution, London, Greater London
  - Local Institution, Belfast
  - Local Institution, Cambridge
  - Local Institution, Cottingham
  - Local Institution, Manchester
  - Local Institution, Tauton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 participants were randomized and treated.
Groups:
- Nivolumab + BMS-986205: Nivolumab 480 mg IV Q4W + BMS-986205 100 mg PO QD
- Nivolumab: Nivolumab 480 mg IV Q4W
Period: Overall Study
Arm/Group | Nivolumab + BMS-986205 | Nivolumab
Started | 10 | 10
Completed | 2 | 1
Not Completed | 8 | 9
Not completed — Disease progression | 4 | 6
Not completed — Study drug toxicity | 1 | 0
Not completed — Participant request to discontinue treatment | 0 | 1
Not completed — Participant withdrew consent | 1 | 0
Not completed — Other reasons | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + BMS-986205 | Nivolumab | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing different types of Adverse Events, including Death, Any cause Adverse Events (AEs), Drug-related AEs, Any cause Serious Adverse Events (SAEs), Drug-related SAEs, SAEs leading to discontinuation, and Drug-related Non-serious AEs leading to discontinuation
Time Frame: From first dose to 30 days following last dose (up to approximately 25 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + BMS-986205 | Nivolumab
Number analyzed (Participants) | 10 | 10
Participants
  Deaths | 0 | 0
  Any cause SAEs (any grade) | 3 | 3
  Drug-related SAEs (any grade) | 1 | 0
  SAEs leading to discontinuation | 1 | 0
  Any cause AEs (any grade) | 10 | 9
  Drug-related AEs (any grade) | 9 | 7
  Drug-Related Non-serious AEs leading to discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to approximately 300 days following last dose. Serious adverse events and non-serious adverse events above 5% were assessed from first dose to 100 days following last dose.
Arm/Group | Nivolumab + BMS-986205 | Nivolumab
All-Cause Mortality (participants affected / at risk) | 1/10 | 3/10
Serious Adverse Events (participants affected / at risk) | 4/10 | 4/10
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + BMS-986205 (N=10) | Nivolumab (N=10)
Constipation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + BMS-986205 (N=10) | Nivolumab (N=10)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Ocular discomfort (Eye disorders) | 0 | 1
Vitreous floaters (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 4
Proctalgia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 5 | 2
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 2
Influenza like illness (General disorders) | 2 | 1
Mucosal inflammation (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Polydipsia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Itching scar (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03329846/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT03329846/SAP_001.pdf